CLINICAL TRIAL: NCT06317064
Title: Diagnostic and Therapeutic Potential of Substance P/ NK1R Receptor in Primary Dysmenorrhea: a Randomized Controlled Trial
Brief Title: Diagnostic and Therapeutic Potential of Substance P/ NK1R Receptor in Primary Dysmenorrhea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lahore Medical Research Center, LLP (Industry)
Responsible Party: Principal Investigator, Riffat Mehboob, Dr., Lahore Medical Research Center, LLP
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LMRC-Aprepitant-Pain-01
Record Dates: First submitted 2024-02-23; First posted 2024-03-19 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-03

CONDITIONS: Primary Dysmenorrhea
Keywords: Substance P; Neurokinin 1 Receptor; Primary Dysmenorrhea; Aprepitant; Rosemary; Ibuprofen
MeSH Terms: interventions — Ibuprofen; Aprepitant; Anti-Inflammatory Agents, Non-Steroidal; Neurokinin-1 Receptor Antagonists

STUDY DESIGN:
Intervention Model Description: Group 1: Controls 10 females with no dysmenorrhea participated as controls. Group 2: NSAIDS All 30 participants in this group used NSAIDs (Non-steroidal Anti-Inflammatory Drugs), during their dysmenorrhea period. Same patients from phase 2 (n=30) in next cycle received NK1R antagonist "Dexamethasone (6mg) + Aprepitant (80mg)" for 2 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): 10 females with no dysmenorrhea participated as controls.
- NSAIDs and Aprepitant group (Sequential) (Experimental): All 30 participants in this group used NSAIDs (Non-steroidal Anti-Inflammatory Drugs), during their dysmenorrhea period. Same patients from phase 2 (n=30) in next cycle received NK1R antagonist "Dexamethasone (6mg) + Aprepitant (80mg)" for 2 days.
  Interventions: Drug: Ibuprofen and Aprepitant

INTERVENTIONS:
Drug: Ibuprofen and Aprepitant — All 30 participants in this group used NSAIDs (Non-steroidal Anti-Inflammatory Drugs), during their dysmenorrhea period. Same patients from phase 2 (n=30) in next cycle received NK1R antagonist "Dexamethasone (6mg) + Aprepitant (80mg)" for 2 days.
  Other Names: NSAIDs, Neurokinin 1 Receptor antagonist
  Arms: NSAIDs and Aprepitant group (Sequential)

SUMMARY:
Dysmenorrhea is characterized as excruciating menstrual cramps of uterine origin and is one of the most prevalent gynecological illnesses. Substance P (SP) and NK1R mediate the symptoms of various pain disorders with chronic and/or neuropathic pain. Objective: To evaluate diagnostic and therapeutic potential of Substance P/ NK1R receptor in primary dysmenorrhea. Study Design: This was a randomized controlled trial which took place at Lahore Medical Research Center from March 2024 to October 2024. Non-probability convenient sampling techniques was used for sampling. A total of 40 female participants was included in the study who met specific criteria for inclusion. The study comprised of three phases, Phase 1 (Before medication), Phase 2 (NSAIDs) and Phase 3(Dexamethasone + Aprepitant). 10 females with no dysmenorrhea participated as controls. The study duration spanned three menstrual cycles. 20 dysmenhorric and 6 controls were analyzed for NK1R levels. Several assessment tools were also used in the study,

DETAILED DESCRIPTION:
This was a randomized controlled trial which took place at Lahore Medical Research Center from March 2024 to October 2024. Non-probability convenient sampling techniques was used for sampling. A total of 40 female participants was included in the study who met specific criteria for inclusion. 10 females with no dysmenorrhea participated as controls. The study duration spanned three menstrual cycles, during which participants were divided into three Phases. Phase 1: Blood samples of all 30 patients were collected prior to any medication. Phase 2: All 30 participants in this phase used NSAIDs (Non-steroidal Anti-Inflammatory Drugs), during their dysmenorrhea period. Phase 3: All the patients from phase 2 (n=30) received NK1R antagonist "Dexamethasone (6mg) + Aprepitant (80mg)" for 2 days. Out of these patients, 20 dysmenhorric and 6 controls were analyzed for NK1R levels.

Data Collection

A 5cc blood sample was collected from each participant on the 2nd day of their menstrual cycle before any intervention. Another 5cc blood sample was collected on the 2nd day of the menstrual cycle after the first intervention. Another 5cc blood sample was collected on the 2nd day of the menstrual cycle after the 2nd intervention. Prior to and following the intervention, a complete blood count (CBC) was conducted to assess any changes in blood parameters. Serum was extracted from the collected blood samples for further analysis.

Human SP and Neurokinin-1 Receptor (NK1R) levels measurement Human SP and its antagonist NK1R levels were analyzed using ELISA technique. This analysis was performed thrice to investigate the role of Substance P and NK1R in menstrual pain before and after the intervention. BT Lab Human Substance P and NK1R ELISA kit was used to measure levels of SP and NK1R in serum samples of participants (Catalogue Numbers: E1528Hu, E6938Hu).

Assessment tools

The study's participants filled out a basic questionnaire meant to collect sociodemographic information and analyze a variety of parameters. Body Mass Index (BMI), Family History of Pain, Age at Menarche, Length of Menstrual Cycle, Age of Onset of Dysmenorrhea, and Sleep Duration were all included in these surveys. The Depression Anxiety Stress Scale (DASS), Visual Analogue Scale (VAS), Mini Nutritional Assessment (MNA), International Physical Activity Questionnaire (IPAQ), and Pictorial Blood Loss Assessment Chart were among the other questionnaires used.

Visual Analogue Scale (VAS)

Female participants' levels of pain were measured using the Visual Analog Scale (VAS). With a scale from 0 to 10, where 10 is the most excruciating pain possible, the VAS is a well-known measure for assessing pain perception. Participants were divided into three groups to reflect varied levels of pain severity based on their VAS ratings obtained throughout the first three consecutive days of both menstrual cycles: Mild Pain, Moderate Pain, and Severe Pain.

Mini Nutritional Assessment (MNA)

The female participants' eating patterns were assessed using the Nestle Nutrition Institute Mini Nutritional Assessment in order to look into any possible associations between their diet and menstrual discomfort. Participants who scored between 24 and 30 had good nutritional status, those who scored from 17 to 23.5 were at risk of malnutrition, and those who scored under 17 were poorly nourished.

Depression Anxiety Stress Scale (DASS-21)

The DASS-21 was used to evaluate the psychological health of our subjects and comprehend how it related to dysmenorrhea. Based on their stated levels of stress, anxiety, and depression, participants were divided into five groups using this scale: normal, mild, moderate, severe, and extremely severe. A score of 0 to 9 indicates normal, 10 to 13 indicates mild depression, 14 to 20 indicates moderate depression, 21 to 27 indicates severe depression, and 28 or above indicates extremely severe depression. Scores between 0 and 7 indicate normal anxiety, 8 to 9 indicate mild anxiety, 10 to 14 indicate moderate anxiety, 15 to 19 indicate severe anxiety, and 20 or more indicate extremely severe anxiety. For stress, 0-14 represents normal, 15-18 represents mild, 19-25 represents moderate, 26-33 represents severe, and 34+ represents really severe stress.

Pictorial Blood Loss Assessment Chart (PBAC)

The Pictorial Blood Loss Assessment Chart (PBAC), a self-administered pictorial assessment chart that assigns scores based on how much tampons and cotton-based sanitary pads stain throughout a menstrual cycle, was given to the patients as a tool to measure their menstrual blood volume [24-26]. Reliability of the PBAC has been shown [25, 26]. They were given guidelines by the researcher on how to utilize the PBAC. Hypomenorrhea was linked to PBAC scores of 10 or less, regular monthly flow was linked to PBAC scores of 10 to 99, and heavy menstrual bleeding was linked to PBAC scores of 100 or more for two months. Cotton pads were the only sanitary goods used. Software for statistical analysis was used to determine scores.

Statistical Analysis

Data analysis was carried out using Graph Pad Prism 8.0.2, a statistical software package. The collected data, including questionnaire responses, CBC results, Substance P and NK1R levels, were analyzed to assess the effects of the interventions on menstrual pain and related factors. Two-way ANOVA test was used for analysis. P-value less than 0.05 was considered significant.

Ethical considerations

This study was approved by Ethical Review Board of Lahore Medical Research Center. The research followed declaration of Helsinki and written and informed consent was taken from all participants.

ELIGIBILITY:
Inclusion Criteria:

The participants must be unmarried women of reproductive age who have moderate to severe dysmenorrhea.

* The participants must experience dysmenorrhea during most menstrual cycles to be included in the study.
* For controls, they must not have dysmenorrhea.

Exclusion Criteria:

Those with irregular or infrequent menstrual cycles.

* Women who are taking oral contraceptive pills (OCPs) and using an intrauterine contraceptive device (IUD) excluded from the study.
* Women who have reached menopause or have undergone a surgical procedure resulting in the cessation of menstruation excluded from the study.
* Women who are pregnant or breastfeeding.
* Women who taking any medication like sedatives and NSAIDs.
* Women with PCOs, hysterectomy and uterine carcinoma will not be included.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — this is study on primary dysmenorrhea, hence all female participants were enrolled
Enrollment: 40 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale Score (Pain scale) | At the end of one cycle (each cycle is of 28-3- days)
  Female participants' levels of pain were measured using the Visual Analog Scale (VAS). With a scale from 0 to 10, where 10 is the most excruciating pain possible, the VAS is a well-known measure for assessing pain perception. Participants were divided into three groups to reflect varied levels of pain severity based on their VAS ratings obtained throughout the first three consecutive days of both menstrual cycles: Mild Pain, Moderate Pain, and Severe Pain
Mini Nutritional Assessment (MNA) Score | At the end of one cycle (each cycle is of 28-3- days)
  The female participants' eating patterns were assessed using the Nestle Nutrition Institute Mini Nutritional Assessment in order to look into any possible associations between their diet and menstrual discomfort. Participants who scored between 24 and 30 had good nutritional status, those who scored from 17 to 23.5 were at risk of malnutrition, and those who scored under 17 were poorly nourished.
DASS-21 (Depression Anxiety Stress Scale) | At the end of one cycle (each cycle is of 28-3- days)
  The DASS-21 was used to evaluate the psychological health of our subjects and comprehend how it related to dysmenorrhea. Based on their stated levels of stress, anxiety, and depression, participants were divided into five groups using this scale: normal, mild, moderate, severe, and extremely severe. A score of 0 to 9 indicates normal, 10 to 13 indicates mild depression, 14 to 20 indicates moderate depression, 21 to 27 indicates severe depression, and 28 or above indicates extremely severe depression. Scores between 0 and 7 indicate normal anxiety, 8 to 9 indicate mild anxiety, 10 to 14 indicate moderate anxiety, 15 to 19 indicate severe anxiety, and 20 or more indicate extremely severe anxiety. For stress, 0-14 represents normal, 15-18 represents mild, 19-25 represents moderate, 26-33 represents severe, and 34+ represents really severe stress.
Pictorial Blood Loss Assessment Chart (PBAC) | At the end of one cycle (each cycle is of 28-3- days)
  The Pictorial Blood Loss Assessment Chart (PBAC), a self-administered pictorial assessment chart that assigns scores based on how much tampons and cotton-based sanitary pads stain throughout a menstrual cycle, was given to the patients as a tool to measure their menstrual blood volume. Reliability of the PBAC has been shown. They were given guidelines by the researcher on how to utilize the PBAC. Hypomenorrhea was linked to PBAC scores of 10 or less, regular monthly flow was linked to PBAC scores of 10 to 99, and heavy menstrual bleeding was linked to PBAC scores of 100 or more for two months. Cotton pads were the only sanitary goods used. Software for statistical analysis was used to determine scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Riffat Mehboob, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No